CLINICAL TRIAL: NCT01377870
Title: Effect and Side Effect of Mesenchymal Stem Cell in Multiple Sclerosis
Brief Title: Evaluation of Autologous Mesenchymal Stem Cell Transplantation (Effects and Side Effects) in Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Royn-nerve-001
Record Dates: First submitted 2011-06-19; First posted 2011-06-21 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2010-08

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis mesenchymal stem cell intravenous injection
MeSH Terms: conditions — Multiple Sclerosis | interventions — Stem Cell Transplantation; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cell free media (Placebo Comparator): 15 patients with relapsing remitting multiple sclerosis who receive cell free media
  Interventions: Biological: injection of cell free media
- mesenchymal stem cell reciepiants (Experimental): Patients with relapsing remitting multiple sclerosis who underwent intravenous injection of mesenchymal stem cells
  Interventions: Biological: intravenous injection of mesenchymal stem cells

INTERVENTIONS:
Biological: intravenous injection of mesenchymal stem cells — 15 patients with relapsing remitting multiple sclerosis underwent intravenous injection of mesenchymal stem cell
  Other Names: stem cell transplantation
  Arms: mesenchymal stem cell reciepiants
Biological: injection of cell free media — Patients who are in control group underwent media injection but after 6 months they will be transplanted by stem cell.
  Other Names: control group
  Arms: cell free media

SUMMARY:
Multiple sclerosis is a multifocal inflammatory disease of the central nervous system which affects young individuals and causes paralysis of the limbs, sensation, visual and sphincter problems. The disease is caused by an autoimmune mechanism, ie the immune system produces antibodies and cells which attack the self myelin antigens, causing therefore demyelination. The disease is clinically evident with relapses of neurological disability due to the dysfunction of the areas (plaques of multiple sclerosis) in which damage of myelin occurs. Disability can accumulate with time and the disease enters a progressive phase due to damage of the axons and irreversible neurodegeneration. Although, effective immunotherapies exist which downregulate the autoimmune anti-myelin reactivity and reduce the rate of relapses of MS (like Copaxone and interferons), there is no effective means today to stop the progression of disability and induce rebuilding of the destroyed myelin.Adult bone marrow derived stromal cells (MSC) were shown to induce similar (to the neuronal stem cells) immunomodulatory and neuroregenerative effects and were shown in our laboratory to induce neuroprotection in the animal model of chronic experimental autoimmune encephalomyelitis (EAE). These bone marrow derived MSCs offer practical advantages for clinical therapeutic applications, since they can be obtained from the adult bone marrow and therefore the patient can be the donor for himself, without any danger for rejection of the cells. In addition, MSCs carry a safer profile and are less prone to malignant transformation.

Our center will perform a clinical trial with intra venous transplantation of bone marrow derived mesenchymal stem cell.our purpose is to evaluate the safety and feasibility of cell transplantation after 1year following up.

DETAILED DESCRIPTION:
In the clinical trial 30 patients with multiple sclerosis who are drug resistance will take apart.Based on inclusion and exclusion criteria patients are chosen.Bone marrow aspiration will be done for all of them under local anesthesia.Patients are randomly divided in 2 groups:case and control. Then mesenchymal stem cells which are separated and prepared will be transplanted by intravenous injection to the patients in case group and the cells which obtain from patients in control group are frozen and inject after 6 months. Patients will be followed by Evaluation of EDSS MSFC RAO Test brain and cervical MRI and quality of life questionnaire after 1th 3th 6th and 12th months after transplantation.all these tests will be done before transplantation as basic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Age: 18-55years
* Duration of disease: 2-10 years
* Relapsing remitting with drug resistance
* EDSS: 3-6.5
* Resistance to immunomodulatory and cytotoxic drugs:

  * At least 1-2 sever relapse during 1 year drug treatment
  * At least increase 1 point of EDSS during 1 year drug treatment
* Secondary progressive or relapsing multiple sclerosis
* Primary progressive MS with relapse or GAD positive enhancement
* Secondary progressive MS with relapse
* Secondary progressive MS without relapse:progression of disease with 1 point increase of EDSS during last 18 months

Exclusion Criteria:

* Pregnancy positive test
* Under treatment with cytotoxic drugs at the same time or during last 3 months
* Under treatment with immunomodulatory drugs at the same time or during last month
* Relapse of disease 30 days or less than 30 days before transplantation
* Primary progressive MS with out relapse or GAD positive enhancement

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-12; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
MRI metrics changes | 6 months
  evaluate the effect of mesenchymal stem cell transplantation on number of GD positive lesions.
Brain atrophy | 12 months
  evaluate the effect of mesenchymal stem cell transplantation to improve brain atrophy
number of sever relapses | 6 months
  evaluation the effect of mesenchymal stem cell transplantation on number of sever relapses
EDSS | 6 months
  Evaluation the effect of mesenchymal stem cells on progression of disease based on EDSS
MSFC | 6 months
  Evaluation the effect of mesenchymal stem cells transplantation on MSFC

SECONDARY OUTCOMES:
quality of life | 6 months
  Evaluation the effect of mesenchymal stem cell transplantation on patients quality of life
RAO Test | 6 months
  Evaluation the effect of mesenchymal stem cell transplantation on RAO Test.
intravenous cell transplantation | 6 months
  evaluation the side effect of intravenous transplantation of mesenchymal stem cell

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of cell therapy center of Royan Institute; Masoud Nabavi, MD, Principal Investigator — scientist and clinician; Leila Arab, MD, Principal Investigator — Department of regenerative medicine,Royan Institute
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://Royaninstitute.org